CLINICAL TRIAL: NCT01933945
Title: OPTIMIS - Outcomes of HCC Patients Treated With TACE Followed or Not Followed by Sorafenib and the Influence of Timing to Initiate Sorafenib
Brief Title: Outcomes of HCC (Hepatocellular Carcinoma) Patients Treated With TACE (Transarterial Chemoembolization) and Early, Not Early or Not at All Followed by Sorafenib
Acronym: OPTIMIS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16560; NX1301 (Other: Company internal)
Record Dates: First submitted 2013-08-29; First posted 2013-09-02 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TACE + early Nexavar: Patients with early start of Sorafenib treatment. This cohort comprises all patients where the physician decides at the time of TACE non-eligibility to choose Sorafenib as the next treatment option (regardless of whether TACE treatment is continued or not).
  Interventions: Procedure: TACE (transarterial chemoembolization); Drug: Sorafenib (Nexavar, BAY43-9006)
- TACE without early Nexavar: Patients without early start of Sorafenib treatment. This cohort comprises all patients where the physician decides at the time of TACE non-eligibility not to choose Sorafenib as the next treatment option. This cohort also includes patients with TACE non-eligibility for whom the decision to treat with Sorafenib is made at a later point in time, patients who are never treated with Sorafenib as well as patients for whom another systemic cancer treatment has been chosen be the physician either at time of TACE non-eligibility or at a later point in time.
  Interventions: Procedure: TACE (transarterial chemoembolization)

INTERVENTIONS:
Procedure: TACE (transarterial chemoembolization) — First treatment for all patients included in the study
Drug: Sorafenib (Nexavar, BAY43-9006)
  Groups: TACE + early Nexavar

SUMMARY:
This study will collect data of patients who are treated with TACE followed by sorafenib for hepatocellular carcinoma (HCC) or patients without Sorafenib after TACE. In contrast to a prior observational study on sorafenib (GIDEON study), where pre-treatment with TACE was documented retrospectively, this study will collect more detailed information about the TACE treatment and the status of a patient when treatment with sorafenib is started.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically/cytologically documented or radiographically diagnosed HCC. Radiographic diagnosis needs typical findings of HCC by radiographic method i.e. on multi-dimensional dynamic CT, CT hepatic arteriography (CTHA)/CT arterial portography (CTAP) or MRI.
* Patients with BCLC (Barcelona clinic liver cancer staging) stage B or higher.
* Patients in whom a decision to treat with TACE has been made at time of study enrollment. Patients that have received one TACE in the past also can be enrolled, if the TACE was done at the same site and all required data about such previous TACEs are available. TACE includes both conventional TACE with lipidiol (or similar agents) and chemotherapeutic agent(s) and TACE with DC Beads excluding TAE without chemotherapeutic agent.
* Patients with unresectable HCC (incurable with curative treatments including resection or ablation or not eligible for resection or local ablation)
* Patients must have signed an informed consent form
* Patients must have a life expectancy of at least 8 weeks

Exclusion Criteria:

* Patients who have received TACE in the past but the data about TACE required in this protocol are not available
* Patients who received any systemic anti-cancer therapy prior to the first TACE
* Patients who are treated according to a trial protocol for intervention including a locoregional therapy or systemic therapy
* Hospice patients
* All contra-indications according to the local marketing authorization should be considered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients with a diagnosis of hepatocellular carcinoma (HCC) will be enrolled in the participating study countries and sites during the enrollment period. All treatment decisions prior inclusion of a patient as well as during the observation must be made by the investigator based on his regular medical practice. Patients must give written informed consent prior to documentation.
  During the course of the study, patients will be assigned to one of the following cohorts of special interest:
  1. Patients with early start of sorafenib treatment
  2. Patients without early start of sorafenib treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1676 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 3 years
  Defined as time (in days) from time of TACE non-eligibility to death due to any cause. Patients lost to follow-up or alive at the end of the study will be censored at the last date known to be alive.

SECONDARY OUTCOMES:
Overall survival from initial TACE | Up to 3 years
  OS from initial TACE was defined as the time interval from the day of the first TACE to death due to any cause.
Progression-free survival (PFS) from initial TACE | Up to 3 years
  PFS from initial TACE was defined as the time interval measured from the day of the first TACE to documented (radiological or clinical) progression or death, whichever came first.
Time to progression (TTP) from initial TACE | Up to 3 years
  TTP from initial TACE was defined as the time interval from the day of first TACE to the date of documented progression.
Tumor response according to mRECIST criteria | Up to 3 years
  Tumor response to TACE by modified Response Evaluation Criteria In Solid Tumors (mRECIST) were evaluated according to the categories "Complete Response", "Partial Response", "Stable Disease", and "Not evaluable" by mRECIST for each TACE.
Duration of TACE treatment | Up to 3 years
  Duration of TACE treatment was defined as the time interval from of the day of first TACE to the date of permanent discontinuation of TACE
Number of patients with TEAEs (treatment emergent adverse events) | Up to 3 years
  Patients were monitored for TEAEs using the NCI-CTCAE Version 4.03.
TACE unsuitability | Up to 3 years
  TACE unsuitability was determined according to selected guidelines
Time to TACE non-eligibility | Up to 3 years
  Determined according to the selected guidelines
Deterioration of liver dysfunction | Up to 3 years
  Deteriorations of liver dysfunction were defined as follow: Deterioration of Child Pugh score (A5, A6, B7, B8, B9); Liver dysfunction reported as AE or deterioration of aspartate aminotransferase, alanine aminotransferase or bilirubin (from Grade 1 to Grade 2-5, from Grade 2 to 3-5, Grade 3 to Grade 4 or 5); Any liver related adverse events or deterioration of liver related events according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03; Change of liver related laboratory data (aspartate aminotransferase, alanine aminotransferase, bilirubin, albumin, prothrombin international normalized ratio [INR])
OS from initiation of sorafenib | Up to 3 years
  OS from initiation of sorafenib was defined as the time interval measured from start date of sorafenib treatment to death due to any cause.
PFS from initiation of sorafenib | Up to 3 years
  PFS from initiation of sorafenib was defined as the time interval measured from the start date of sorafenib treatment to documented (radiological or clinical) progression or death, whichever came first.
Tumor status at different visits response according to mRECIST | Up to 3 years
  mRECIST: modified Response Evaluation Criteria In Solid Tumors
Duration of sorafenib treatment | Up to 3 years
  Duration of sorafenib treatment was defined as the time interval from start date of sorafenib treatment to the date of permanent discontinuation of sorafenib treatment (regardless of the reason for discontinuation including death).
TTP from initiation of sorafenib | Up to 3 years
  TTP from initiation of sorafenib was defined as the time interval from start date of sorafenib treatment to the date of documented progression.

OTHER OUTCOMES:
PFS from TACE non-eligibility | Up to 3 years
  PFS from TACE non-eligibility was defined as the time interval from TACE non-eligibility to documented (radiological or clinical) progression or death, whichever came first.
TTP from TACE non-eligibility | Up to 3 years
  TTP from TACE non-eligibility was defined as the time interval from TACE non-eligibility to the date of documented progression.
Tumor response from time of TACE non-eligibility by mRECIST | Up 3 years
  Planned to be evaluated according to the categories "Complete Response", "Partial Response", "Stable Disease", and "Not evaluable"
Switch to sorafenib or other systemic and non-systemic cancer therapy | Up to 3 years
  Evaluated according to the categories "Before initial TACE", "After one TACE", "After two TACEs", and "After more than two TACEs"
Deviations from recommendations for TACE use | Up to 3 years
  Deviations from recommendations for TACE use in the treatment guidelines for TACE use based on the number of patients for whom the treatment decision for a new TACE was made by the investigator after TACE non-eligibility.
Duration of treatment of sorafenib after TACE | Up to 3 years
  Defined as days from the first sorafenib dose to the date of permanent discontinuation of sorafenib plus one

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (31):
- Multiple Locations, Austria
- Multiple Locations, Brazil
- Multiple Locations, Canada
- Multiple Locations, China
- Multiple Locations, Czechia
- Multiple Locations, Denmark
- Multiple Locations, Egypt
- Multiple Locations, France
- Multiple Locations, Greece
- Multiple Locations, Hong Kong
- Multiple Locations, Hungary
- Multiple Locations, India
- Multiple Locations, Indonesia
- Multiple Locations, Israel
- Multiple Locations, Japan
- Multiple Locations, Kazakhstan
- Multiple Locations, Mexico
- Multiple Locations, Netherlands
- Multiple Locations, Pakistan
- Multiple Locations, Poland
- Multiple Locations, Russia
- Multiple Locations, Singapore
- Multiple Locations, Slovakia
- Multiple Locations, South Korea
- Multiple Locations, Spain
- Multiple Locations, Sweden
- Multiple Locations, Switzerland
- Multiple Locations, Taiwan
- Multiple Locations, Thailand
- Multiple Locations, Turkey (Türkiye)
- Multiple Locations, Vietnam